CLINICAL TRIAL: NCT06517368
Title: Ultrasound Elastography Combined With Conventional MRI in Differentiating Solid Renal Parenchyma Masses
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Mohamed Sayed, Resident, Assiut University
Other Study IDs: renal masses
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Renal Masses
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign solid renal masses
  Interventions: Device: MRI, Ultrasound
- malignant solid renal masses
  Interventions: Device: MRI, Ultrasound

INTERVENTIONS:
Device: MRI, Ultrasound — The patients will undergo both B-mode and sonoelastographic examinations in the supine and lateral decubitus position and will perform during breath-holding after deep inspiration. The elastogram was displayed over the B-mode image in a color scale: red (greatest strain, softest tissue component), green (average strain, intermediate tissue component), and blue (no strain, hardest tissue component) Patients will be examined by MRI with diffusion images and ADC values.

SUMMARY:
Investigate the diagnostic accuracy of Ultrasound Elastography combined with conventional MRI in evaluation of solid renal masses using histopathology as a gold standard.

DETAILED DESCRIPTION:
Renal masses are increasingly detected incidentally during imaging that plays a key role in the characterization of these masses. Renal masses are a biologically heterogeneous group of tumors ranging from benign masses to cancers that can be indolent or aggressive.Typical imaging methods available for differentiating benign from malignant renal lesions include ultrasound (US), contrast-enhanced ultrasound (CEUS), computed tomography (CT), and magnetic resonance imaging (MRI). Renal mass biopsy is considered the gold standard for determining the presurgical histology of renal masses. US can easily characterize most incidental renal masses , but it cannot always differentiate between benign and malignant solid renal tumors.MR imaging has been gaining popularity in recent years as a problem-solving tool in the evaluation of renal masses.It has several advantages including no exposure to radiation and a superior soft-tissue contrast, and may be a feasible initial imaging option for characterization of renal tumors.Ultrasound elastography (USE) is an imaging technology sensitive to tissue stiffness that was first described in the 1990s.It takes advantage of the changed elasticity of soft tissues resulting from specific pathological or physiological processes. Ultrasound-based methods include strain elastography, two-dimensional shear wave elastography (2D-SWE), point shear wave elastography (pSWE), and vibration-controlled transient elastography (VCTE). US elastography is a non-invasive technique that can assess tissue elasticity, has shown promising results in many clinical settings, and could be able to differentiate between benign and malignant renal lesions based on tissue stiffness.

ELIGIBILITY:
Inclusion Criteria:

* patient with solid renal masses.

Exclusion Criteria:

* patient with cystic renal masses.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients will undergo both B-mode and sonoelastographic examinations in the supine and lateral decubitus position and will perform during breath-holding after deep inspiration. The elastogram was displayed over the B-mode image in a color scale: red (greatest strain, softest tissue component), green (average strain, intermediate tissue component), and blue (no strain, hardest tissue component) Patients will be examined by MRI with diffusion images and ADC values.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Elastography combined with conventional mri in differentiating solid renal parenchyma masses | Baseline
  Investigate the diagnostic accuracy of Ultrasound Elastography combined with conventional MRI in evaluation of solid renal masses using histopathology as a gold stsndard.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt